CLINICAL TRIAL: NCT04694898
Title: Integrating Health and Agriculture Services for Improved Household Food Security and Nutritional Status of Mothers and Children 4-6 Years of Age
Brief Title: Sustainable Undernutrition Reduction in Ethiopia
Acronym: SURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Ethiopian Public Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-08862
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2020-12

CONDITIONS: Stunting; Dietary Deficiency; Anemia
Keywords: Stunting; Diet diversity; Food production; Household food security; Women empowerment; Knowledge, Attitudes and Practices; Anemia; Malaria
MeSH Terms: conditions — Growth Disorders; Malnutrition; Anemia; Behavior; Malaria | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study is part of the evaluation of the Government project "SURE". SURE intervention districts were pre-selected in four regions out of the nine regions in Ethiopia. The regions were selected because they are agrarian and have high food insecurity and stunting prevalence (Oromia, Amhara, SNNPR and Tigray). A total of 36 districts were selected and assigned to the SURE intervention.
  Comparison control districts were selected in equal number in the same four agrarian regional strata. Districts were roughly matched based on stunting prevalence tertiles (low, medium or high) and food insecurity scores. Eligible households are households with at least one child under the age of 2 years. The intervention started in 2016 and included 4299 households, 2146 of which were included in the intervention group and 2153 in the control group. After baseline data collection, all households in the intervention group received counselling at household and community levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Households in the control arm receive standard/national nutrition specific interventions, i.e. growth monitoring, vaccination, vitamin A supplementation and deworming
  Interventions: Behavioral: Standard programme
- SURE Intervention (Experimental): Households in the intervention group with children younger than 2 years benefit from:
  1. Interpersonal contacts to provide counselling on infant and young child feeding practices (IYCF) and nutrition-sensitive agriculture advice to mothers and fathers of children under 24 months, inclusive of pregnant women and fathers-to-be, jointly delivered by the local health and agriculture extension workers during routine household visits
  2. Men's and women's group dialogues targeting all men and women in a given community network, facilitated also by the local health and agriculture extension workers
  3. Media campaign to reinforce IYCF and dietary diversity messages
  Interventions: Behavioral: SURE intervention

INTERVENTIONS:
Behavioral: Standard programme — The control arm will receive national standard programme for women and children under the age of 2 years. This includes 1) national nutrition and health care including iron & folic acid (IFA) supplementation in pregnancy; 2) early initiation and exclusive breastfeeding until 6 months of age; 3) timely introduction of liquid and semi-solid complementary foods; and 4) diversified complementary foods.
  Other Names: Control
  Arms: Control
Behavioral: SURE intervention — The SURE package includes: 1) promoting diversified agriculture; 2) promoting infant and young child feeding practices; 3) women empowerment in decision making related to agriculture, food and health; and 4) enhanced food security and Water, Sanitation and Hygiene ("WASH") practices.
  Other Names: Intervention
  Arms: SURE Intervention

SUMMARY:
The causes of malnutrition are complex and addressing the problem requires integrated action among various sectors. Globally, much attention has been given to nutrition-specific interventions to address the immediate causes of undernutrition. But undernutrition prevalence is decreasing at a very slow rate. Nutrition-specific interventions address the immediate determinants of child undernutrition, such as inadequate food and nutrient intake, but do not consider the underlying causes such as food insecurity, poverty, and limited access to clean water, hygienic environments, and health services.

Ethiopia still has a high prevalence of undernutrition. The current situation of food insecurity and malnutrition in Ethiopia has pressurized the government in pursuing a number of nutritional-sensitive interventions to increase diversified food production and consumption like the Sustainable Undernutrition Reduction Program (SURE).

This study aims to investigate whether joint nutrition specific and sensitive interventions can lead to improved household food security, dietary diversification and improved nutritional status in Ethiopian mothers and their young children.

The study will be a community based longitudinal design and will use multistage cluster sampling at the Kebele and household levels in Amhara, Oromia, and Southern Nations, Nationalities, and Peoples' Region (SNNPR) regions.

Households will be randomly selected from the intervention and the non-intervention arms at Kebele level, with 15 households per Kebele. The same children whose baseline are available who were 0-23 months of age at the time of the baseline assessment in 2016 will be recruited as well as their mothers. This represents approximately third of the total sample size at baseline.

DETAILED DESCRIPTION:
Globally 25% of children under age 5 years of age are stunted, i.e. the child's height is more than 2 standard deviations (SD) below the median length/height-for-age as determined by the world health organization child growth standards. Sub-Saharan Africa remains the region with the highest prevalence of undernutrition. Stunting, a multifactorial condition, develops as a result of sustained inadequate nutrition and recurrent infections. Socioeconomic and environmental factors are considered to be important determinants of stunting. Stunting has long term detrimental effects on cognitive development, school achievement and income and hence potentially perpetuates the vicious circle of poverty and malnutrition. Interventions that target directly maternal and child health and nutrition such as maternal supplementation with iron and folic acid and promotion of exclusive and continued breastfeeding, have proven effective in enhancing child and maternal nutrition status and in reducing mortality in women and children. The evidence accumulated over the previous years has also shown that if nutrition-sensitive approaches (i.e. women's empowerment, agriculture, food systems and education) are integrated in nutritional-specific interventions, they can significantly accelerate progress in countries with the highest burden of maternal and child undernutrition and mortality.

Diversified diet provides a balance of nutrients that promote healthy growth and development. Agricultural interventions to improve production of micronutrient-rich foods, through increased productivity, home gardening and diversification efforts have a significant potential to improve dietary diversity and micronutrient intake of children. However, in Ethiopia there is limited evidence on the contribution of nutrition-sensitive agricultural interventions on dietary diversity and nutritional status of children. Our study evaluates a larger governmental programme "sustainable undernutrition reduction in Ethiopia (SURE)", a multi-sector integrated health and agriculture programme that aims to strengthen the existing nutrition specific interventions by addressing two key determinants of undernutrition: inadequate complementary feeding and household dietary diversity.

The SURE package includes: 1) promoting diversified agriculture; 2) promoting infant and young child feeding practices; 3) women empowerment in decision making related to agriculture, food and health; and 4) enhanced food security and Water, Sanitation and Hygiene (so-called "WASH") practices.

The programme started in 2016 and is implemented by the Ministries of Health and Agriculture in Ethiopia through a funding by the Children's Investment Fund Foundation (CIFF). The Ethiopian Public Health Institute (EPHI) has been contracted by the Ethiopian Ministry of health to deliver the programme and to carry out its evaluation at the level of impact, process and cost-effectiveness.

Aims of the Study The study aims to investigate whether access to diversified food through improved nutrition education and enhanced diversity in local and household food production leads to improved household food security, which in turn results in diversified dietary consumption and improved nutritional status of children 4 -6 years of age.

In a control longitudinal study design, our primary objective is to assess the extent of diversified food production and consumption as a result of SURE intervention and to evaluate their effects on nutritional status of children in the target/intervention communities compared to the agricultural practices, food insecurity and nutritional status of children in comparable communities in the control group.

Our second objective is to identify factors that mediate the association between diversified food production and diversified food consumption and design a model for a modified intervention to strengthen the association between diversified food production and consumption at a household level.

Our third objective is to identify key barriers and opportunities of adopting infant and young child feeding practices (IYCF) and nutrition sensitive agriculture interventions.

Methodology The study is part of the evaluation of the government project "SURE". The evaluation will have a mixed-method study design (quantitative and qualitative). A longitudinal survey will be carried out in a representative sample of households four years post-intervention, at the end 2020. The survey will use multistage cluster sampling at the Kebele and household levels.

Quantitative data

Baseline data collection: The survey at baseline collects data on: 1) child (6-23 months) nutritional status (height, weight, and hemoglobin concentration); 2) Infant and YCF practices including breastfeeding, minimum meal frequency, minimum dietary diversity and minimum acceptable diet; 3) maternal knowledge, attitude and practice regarding IYCF; 4) women empowerment; 5) household food insecurity and dietary diversity; 6) water, sanitation and hygiene (WASH); and 7) health services and morbidity symptoms of the child during the 15 day-preceding the interview day (received vitamin A supplement in the previous 6 months; diarrhea; cough; fever and; attending the growth monitoring program).

Key behaviors and agriculture outcomes at household level in the intervention and in the control groups will also be collected. These are: number of trainings organized in the community; crop production diversity; animal husbandry (eggs, chicken, milk, small and large livestock for meat).

In addition to outcome indicators, socioeconomic indicators such as age, ethnic group and education level will also be collected.

Follow-up data collection: follow-up surveys will be conducted after an exposure of four years in the intervention and the control groups. The same indicators collected at baseline will be collected during 2020 but in households with children who will now be 4-6 years of age (hypothetically these children would have been exposed to the intervention).

Qualitative data Qualitative methods will be used to examine the quality of implementation mechanisms of change, and contextual data to help interpret findings of the impact evaluation. Additionally, household expenditure will be estimated to determine the average cost of the intervention per case of stunting averted

ELIGIBILITY:
Inclusion Criteria:

* Children 4 years - 6 years and their mothers/fathers and caregivers
* Participated in the baseline survey (2016)
* Resided in the Control communities during the last four years (control arm), or in the SURE intervention communities (intervention arm).

Exclusion Criteria:

-

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1292 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (g/dl) | Changes in hemoglobin (g/dl) and in prevalence of anemia (<11g/dl) will be measured over the course of the four year program period.
  Hemoglobin concentrations (g/dL)
Linear growth (Z-score and prevalence) | Change in height-for-age Z-scores will be measured as well as the change in the prevalence of stunting (HAZ<-2) over the course of the four year program period.
  Child height (cm) and its Z-score

SECONDARY OUTCOMES:
Dietary diversity (%) | Baseline (2016) and after 4 years at endline (2020)
  Measured with a questionnaire using a qualitative food frequency questionnaire. Unit: Number of food group consumed and percentage of children having consumed 4 groups (upon 7) the previous three days.
Food insecurity access prevalence (%) | Baseline (2016) and after 4 years at endline (2020)
  Measured with a questionnaire to calculate the Household Food Insecurity Access score.
Women's empowerment in agriculture (%) | After 4 years of intervention (endline, 2020)
  Measured by questionnaire, It measures the roles and extent of women's engagement in the agriculture sector in five domains: (1) decisions about agricultural production, (2) access to and decision making power over productive resources, (3) control over use of income, (4) leadership in the community, and (5) time use. Percentage of women over a calculated score.
Maternal knowledge of child care practices related to health/diet/WASH (%) | Baseline (2016) and after 4 years at endline (2020)
  Using questionnaire on knowledge. Percentage of women giving adequate answer.
Maternal practices of child care related to health/diet/WASH (%) | Baseline (2016) and after 4 years at endline (2020)
  Using questionnaire on practices. Percentage of women giving adequate answer.
Child weight (Z-score and %) | Measurements were made for children between the ages of 0 and 23 months of age at baseline and 4 years later, at endline, when the children are between the ages of 4 and 6 years.
  Child weight (kg) and its Z-score
Agricultural production diversity | Baseline (2016) and after 4 years at endline (2020)
  The production of different food groups by the household members that correspond to those groups used in the dietary diversity index.

OTHER OUTCOMES:
Wasting (Z-score and %) | Baseline in children 0-23 months of age and endline in children 4-6 years of age
  Child weight for height Z-score

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent
Locations (1):
- Ethiopia Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
All the data collected in the evaluation survey will be used in the analyses and shared as necessary.

REFERENCES:
- [Result] Ruel MT, Alderman H; Maternal and Child Nutrition Study Group. Nutrition-sensitive interventions and programmes: how can they help to accelerate progress in improving maternal and child nutrition? Lancet. 2013 Aug 10;382(9891):536-51. doi: 10.1016/S0140-6736(13)60843-0. Epub 2013 Jun 6. PMID 23746780
- [Result] Reinbott A, Schelling A, Kuchenbecker J, Jeremias T, Russell I, Kevanna O, Krawinkel MB, Jordan I. Nutrition education linked to agricultural interventions improved child dietary diversity in rural Cambodia. Br J Nutr. 2016 Oct;116(8):1457-1468. doi: 10.1017/S0007114516003433. Epub 2016 Oct 5. PMID 27702425
- [Result] Bahru BA, Jebena MG, Birner R, Zeller M. Impact of Ethiopia's productive safety net program on household food security and child nutrition: A marginal structural modeling approach. SSM Popul Health. 2020 Aug 26;12:100660. doi: 10.1016/j.ssmph.2020.100660. eCollection 2020 Dec. PMID 33005722
- See also: Creating Homestead Agriculture for Nutrition and Gender Equity (CHANGE) in Burkina Faso (CHANGE) — https://clinicaltrials.gov/ct2/show/study/NCT02236468